CLINICAL TRIAL: NCT06042023
Title: REmote Monitoring for preOperaTive Risk assEssment for Major Abdominal Surgery
Brief Title: Remote Patient Monitoring for Preoperative Risk Assessment
Acronym: REMOTES
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Leeds (Other)
Collaborators: The Leeds Teaching Hospitals NHS Trust (Other)
Responsible Party: Principal Investigator, David Jayne, Professor of Surgery, University of Leeds
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: GS22/148530
Record Dates: First submitted 2023-09-04; First posted 2023-09-18 (Actual); Last update posted 2023-09-18 (Actual); Status verified 2023-09

CONDITIONS: Abdominal Neoplasm; Surgery; Surgery-Complications; Risk Assessment
MeSH Terms: conditions — Abdominal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Remote monitoring (Experimental): Participants that consent to the study will undergo additional remote monitoring with the applied wearable sensor.
  Interventions: Device: Lifesignals Wearable Sensor

INTERVENTIONS:
Device: Lifesignals Wearable Sensor — The participants will wear the patch for 3-5 days and be provided with the mobile device, which records data transmitted wirelessly directly from the biosensor patch. During the monitoring period, participants can continue their normal activities.
  Remote monitoring will be undertaken using the CE-marked LifeSignals wearable biosensor. The biosensor communicates with a commercially available mobile device, which relays data to a secure Cloud server (GDPR compliant data transfer).
  Participants will subsequently undergo their planned surgery in the usual way. Data captured from the remote monitoring will not be used or made accessible to inform decisions about clinical care.
  There will be no clinical intervention from the researchers if abnormalities in vital signs are picked up by the monitoring patch, as all data will be analysed retrospectively after the participant's operation. Any clinical concerns about the device that arise will be reported to the relevant clinical team.

SUMMARY:
Preoperative risk assessment (an evaluation of overall health before surgery) is important to determine the overall risk of mortality and complications for patients undergoing major abdominal surgery to allow the appropriate allocation of sparse hospital resources. The current gold standard for preoperative assessment is cardiopulmonary exercise testing (CPET). CPET is, however, not available in all centres that perform major surgery, it is a costly test, and therefore only high-risk patients are tested. Finding new ways of conducting preoperative assessment could improve overall surgical safety, patient experience and reduce cost.

The preoperative use of remote vital signs monitoring can provide important information about the patients' fitness and overall health and may be used for preoperative assessment. This study will use a remote monitoring patch to monitor patients' vital signs before surgery. The aim is to evaluate the utility and patient acceptability of the remote monitoring system and the feasibility of a randomised controlled trial of this type of assessment. Additionally, the study will assess the correlation between the data captured by the remote monitoring system and the CPET results to evaluate the remote monitoring system's ability to predict risk of surgery.

The study will take place in Leeds Teaching hospitals. Adult patients undergoing major abdominal surgery that require CPET before surgery are eligible. Participants will be monitored at home with the patch monitor for 3-5 days before surgery, in addition to their planned preoperative assessment. During remote monitoring, patients will be asked to complete questionnaires on their general health and experience using the patch paired with the mobile phone as part of the monitoring system. Clinical data from the electronic hospital records and general practitioner records available on the trust system will then be collected after surgery to assess complications and calculate risk scores.

DETAILED DESCRIPTION:
The clinical research team will identify eligible participants from standard CPET booking forms, which are received 1 - 2 weeks prior to the test. Researchers involved in this single centre study are part of the clinical care team and have routine access to patient identifiable information. Participants fulfilling the eligibility criteria will be sent a Patient Information Sheet (PIS) explaining the study to accompany the routine appointment letter. Participants attending their CPET appointment will be approached for inclusion in the study by the clinical research team. Participants willing to take part in the study will be asked to provide written, informed consent. CPET will be undertaken in the usual manner, after which the patient will be fitted with a wearable patch and trained to use the remote monitoring software/mobile device. A dedicated mobile device will be provided for the duration of the remote monitoring and returned when the patient is admitted for surgery.

The participants will wear the patch for 3 to 5 days and be provided with the mobile device (modified smartphone), which records data transmitted wirelessly directly from the biosensor patch. During the monitoring period, participants can continue their normal activities as usual. The patch is water resistant, so participants can shower and pat dry the patch with a towel.

The system (patch - mobile device) is reliable and secure, using robust Wi-Fi radio encryption and GDPR (General Data Protection Regulation) compliant data transfer to a separate cloud server. The device cannot be used as a regular phone to make phone calls/browse the web. In the unfortunate event that a device gets lost/ broken, or stolen, the participant will not be liable.

Remote monitoring will be undertaken using the LifeSignals wearable biosensor (www.LifeSignals.com) and the Asclepius software platform. The biosensor communicates with a commercially available mobile device, which relays data to a secure Cloud server. The biosensor is CE-marked and has been used in other clinical settings for remote patient monitoring. The device is currently not routinely used in the NHS.

Participants will subsequently undergo their planned surgery in the usual way. Data captured from the remote monitoring will not be used or made accessible to inform decisions about clinical care.

All decisions regarding perioperative care will be based on the standard preoperative assessment per routine care. The remote monitoring data will not be monitored in real-time. There will be no clinical intervention from the researchers if abnormalities in vital signs are picked up by the monitoring patch, as all data will be analysed retrospectively 90 days after the participant's operation. Any clinical concerns about the device that arise will be reported to the relevant clinical team. In the unlikely event that patient safety is considered at risk in any way as a result of the study intervention, the patient will be withdrawn from the study, and the clinical team and Chief Investigator will be notified, who will escalate the concern to the Sponsor as necessary. The Sponsor or Chief Investigator may take appropriate safety measures to protect research participants against any immediate hazard to their health or safety. In the event of a safety breach, the main REC will be notified within three days on why such measures have been taken. Any other unexpected events will be reported to the REC within 15 days of the research team becoming aware and to the Sponsor within one working day.

Interviews The investigators aim to interview both main study participants and non-participants (CPET only group). Participants fulfilling the eligibility criteria for the main study will be sent an additional Interview Patient Information Sheet to accompany the main study PIS and the routine appointment letter. The approach will take place at the scheduled CPET appointment. A purposive approach to sampling will be used, accounting for age, sex, ethnicity, indication for surgery, and type of surgery. A maximum of 20 study participants and 5 non-participants will be interviewed. Main study participants will be invited to keep a diary of their experiences with the device. For this group, the interview will be scheduled after discharge from the hospital when convenient for the participant.

For the CPET-only group, the timing of the interview will coincide with the timing of approach at the CPET appointment.

The interviews will be semi-structured and last 30-60 min. They will be facilitated by telephone or face-to-face according to the current guidelines on social distancing, investigating participants' attitudes and experiences with the device or what reasons have influenced their decision to decline participation.

The investigators also aim to interview clinicians who are considered to be opinion holders. The participants will be employed by Leeds Teaching Hospitals Trust and will also be provided with a PIS and asked to sign an informed consent form. Again the interview will be facilitated by telephone or face-to-face according to the current guidelines on social distancing, when convenient for the clinician. The interviews will be semi-structured, last 30-60 min, and investigate clinicians' attitudes towards the device.

All interviews will be audio recorded and transcribed verbatim for content analysis.

Data management

Data collection during the study will be handled in accordance with Data Protection Act 2018. An agreement will be in place between the University of Leeds and Asclepius for the provision of the biosensor patches and mobile phones and to cover data transfer, storage, and processing. All information collected will be kept strictly confidential. Information will be held securely on paper and/or electronically at Leeds Teaching Hospitals NHS Trust. A site file and study master file will be held securely within the Clinical Research Office at St James's University Hospital. The study master file will contain all participant information, including the contact information for potential participants from the clinical teams, consent forms, and copies of completed case report forms (CRFs) for the study.

Data collected during the monitoring period will be filtered, compressed, and encrypted, converting analogue biological sensor data to a digital format using the global standard of Advanced Encryption Standard (AES) protocol. The data is then instantly communicated to a central server in a pseudo-anonymised format and is password protected. No patient identifiable data will be entered into the Asclepius platform. The Asclepius cloud database system adheres to all hospital security procedures and data backup policies. At the end of the study, the collected data (monitoring data and questionnaire responses) will be downloaded and consequently erased from the cloud database. All downloaded data will be entered into a secure, password-protected study database on University of Leeds computers within the trust clinical research office. Only the clinical research team will have access to the stored data. Information to link participant numbers and patch numbers to personal data will be kept safely on paper in the study master file in the clinical research office at St James's University Hospital. This information will not be stored in any other way. The trial data will be securely archived for a minimum of 5 years at the end of the study, in accordance with the Good Clinical Practice guidelines.

If a participant withdraws, all data collected by the patch up to that point will be retained unless they explicitly withdraw consent. In the unlikely event that, during the study, a participant loses capacity, any intervention outside of standard care (such as the monitoring patch) will be removed. No further information will be collected after this point in time. Information collected previously to this will remain in the study.

Audio recordings The electronic voice recordings will be transcribed by the research team for content analysis (within three months from the interview), with personal details censored to ensure anonymity (unique study ID). The investigators will only store these recordings for as long as necessary on a secure University of Leeds server. The audio file will be deleted permanently immediately after the recording gets transcribed. The transcribed recordings will then be stored securely for 5 years on the University of Leeds servers before being permanently deleted.

With regards to the analysis of the interview content, a thematic framework approach to analysing data will be used. This approach is widely used in applied health research. There are five stages of data analysis summarised below:

I) familiarisation with data; II) identifying a thematic framework; III) indexing; IV) charting; and V) mapping and interpretation

The process enables the researcher to identify emerging themes in the data. The thematic analysis will be modified in light of new data, and a process of iterative comparison will be used to examine across themes and cases, capturing the participant experience of being part of the study and using the device.

Participants are free to withdraw from the substudy up to 7 days after the interview. After this time, transcriptions will be anonymised, and it may not be possible to identify the participant. It is possible to withdraw from the optional study and continue in the main study. The investigators will still keep records from the interview unless the participant explicitly withdraws consent for this. In the unlikely event that, during the study, the participant loses capacity, any intervention outside of standard care (for main study participants) will be removed. No further information will be collected after this point in time. Information collected previously to this will remain in the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing elective major abdominal surgery (BUPA classification: Major 1 to +5) [36]
* Patients who can be trained to use the remote monitoring software on a dedicated smartphone
* Patients who have the capacity to provide informed, written consent
* Patients referred for CPET as part of routine preoperative assessment
* Ages ≥ 18 years
* Patients who can comprehend verbal and written English

Exclusion Criteria:

* Patients allergic to skin adhesive
* Patients with a cardiac pacemaker
* Patients who do not need to undergo CPET for preoperative assessment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2022-12-19 (Actual); Primary Completion 2024-06-19 (Estimated); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
Recruitment rates | up to 18 months
  Ratio of patients recruited in the study to overall number of eligible patients approached
Utility as measured by the System Usability Questionnaires. | up to 18 months
  Will be assessed with System Usability score questionnaires filled by participants

SECONDARY OUTCOMES:
Acceptability of the Remote monitoring system as evidenced by qualitative interviews. | up to 18 months
  Patients are invited to take part in an interview process if they are willing to elaborate and provide their thoughts and experiences on the system.
  In addition all patients fill in specific questionnaire regarding their experience of the remote monitoring system at the end of the monitoring process.
Number of Predictors extracted from the wearable data. | up to 21 months
  Feature extraction and machine learning analysis of the wearable raw data will determine which predictors might be significant during the development of a predictive model process. (Such predictors might include factors such as Heart rate, Heart rate variability, Heart rate reserve, foot step count, walking distance, walking speed, respiratory rate).

CONTACTS AND LOCATIONS:
Overall Officials: Alexios Dosis, MD, Principal Investigator — Leeds institute of Medical Research
Locations (1):
- Leeds Teaching Hospitals, Leeds, United Kingdom